CLINICAL TRIAL: NCT00084110
Title: Complementary Alternative Medicine
Brief Title: Use of Complementary and Alternative Medicine Among Older Mexican Americans
Status: Terminated | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: K08AT000722-03 (NIH)
Record Dates: First submitted 2004-06-07; First posted 2004-06-08 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Arthritis; Diabetes Mellitus; Fractures; Hypertension; Depression; Urinary Incontinence
Keywords: Aged; Mexican Americans; Complementary Therapies
MeSH Terms: conditions — Arthritis; Diabetes Mellitus; Fractures, Bone; Hypertension; Depression; Urinary Incontinence

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to examine complementary and alternative medicine use among older Mexican Americans and to determine how this use influences physical, functional, and mental health.

DETAILED DESCRIPTION:
Alternative medicine has received increasing attention from both the scientific and public communities. While the majority of current alternative medicine use is the result of interest in replacing or augmenting formal medical treatments, several cultures have long-standing traditions of herbal medicine use, particularly among older, more traditional members. Research in this area has been limited primarily to small-scale studies that identify herbal remedies popular in specific cultures. This study observes older Mexican Americans because a substantial proportion of this population continue to utilize traditional herbal remedies in their everyday life.

ELIGIBILITY:
Inclusion Criteria:

* Mexican American

Exclusion Criteria:

* Unable to complete survey questionnaire

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 3000
Dates: Start 1993-08; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- Jose A. Loera, Galveston, Texas, United States

REFERENCES:
- [Background] Loera JA, Black SA, Markides KS, Espino DV, Goodwin JS. The use of herbal medicine by older Mexican Americans. J Gerontol A Biol Sci Med Sci. 2001 Nov;56(11):M714-8. doi: 10.1093/gerona/56.11.m714. PMID 11682580